CLINICAL TRIAL: NCT02293200
Title: TWO METHODS OF TRAINING TO IMPROVE CHEST COMPRESSION EFFECITVENESS BY MEDICAL STUDENTS AND BYSTANDERS: A Randomized Trial
Brief Title: CPR Feedback Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPR/2014/03
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional learning (Experimental): chest compression group learning without CPR feedback device. After a month of quality control of chest compressions is made also without the device.
  Interventions: Device: Standard BLS
- Experimental learning (Experimental): Training is done using TrueCPR feedback device. After a month of quality control of chest compressions is made without the device. To do this will be indicated on the impact of the use of feedback devices for improving the effectiveness of training in CPR.
  Interventions: Device: Standard BLS; Device: TrueCPR

INTERVENTIONS:
Device: Standard BLS — basic life support without any feedback device
Device: TrueCPR — CPR with feedback device
  Arms: Experimental learning

SUMMARY:
The aim of the study was to compare two methods of training in CPR, standard basic life support and CPR using CPR feedback device.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study

Exclusion Criteria:

* Not meet the above criteria
* Wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Effective compressions compression with correct depth (40-50mm), correct hand position and complete decompressions | 1 month
  effective compressions was defined as compression with correct depth (40-50mm), correct hand position and complete decompressions

SECONDARY OUTCOMES:
effective compressions ratio effective compressions [%] multiplied by flow time [%] | 1 month
  effective compressions ratio was defined as effective compressions [%] multiplied by flow time [%]
Flow time sum of all periods during which chest compressions were performed. | 1 month
  flow time was defined as the sum of all periods during which chest compressions were performed.
absolute hands-off time sum of all periods without chest compressions or ventilation | 1 month
  absolute hands-off time (HOT) was defined as the sum of all periods without chest compressions or ventilation
Compression depth compression in correct depth (40-50mm) measured by the software is connected to the manikin and computer | 1 month
  compression in correct depth (40-50mm) measured by the software is connected to the manikin and computer

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland